CLINICAL TRIAL: NCT00566618
Title: Phase I/II Study of Dasatinib in Combination With Zoledronic Acid for the Treatment of Breast Cancer With Bone Metastasis
Brief Title: Dasatinib in Combination With Zoledronic Acid for the Treatment of Breast Cancer With Bone Metastasis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0900; NCI-2015-01920 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-11-29; First posted 2007-12-03 (Estimated); Results first posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Breast Cancer; Bone Metastases
Keywords: Breast Cancer; Bone Metastases; Breast Cancer with Bone Metastases; Breast Cancer with Metastases to Bone; Dasatinib; Zometa; Zoledronic Acid; Zoledronate; BMS-345825; Sprycel®
MeSH Terms: conditions — Breast Neoplasms | interventions — Dasatinib; Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dasatinib + Zoledronic Acid (Experimental): Dasatinib Phase I: First Cohort = 100 mg PO Daily x 28 days; Next Cohort = Dose Expansion or Reduction Based on Dose Limiting Toxicity (DLT) in Initial Cohort.
  Zoledronic Acid Phase I: First Cohort = 4 mg IV Over 15 min. every 4 Weeks; Next Cohort = Dose Expansion or Reduction Based on Dose Limiting Toxicity (DLT) in Initial Cohort. Phase II: Recommended Phase II Dose (RP2D) as determined with Phase I.
  Interventions: Drug: Dasatinib; Drug: Zoledronic Acid

INTERVENTIONS:
Drug: Dasatinib — Phase I: First Cohort = 100 mg PO Daily x 28 days; Next Cohort = Dose Expansion or Reduction Based on Dose Limiting Toxicity (DLT) in Initial Cohort.
  Phase II: Recommended Phase II Dose (RP2D) as determined with Phase I.
  Other Names: BMS-345825; Sprycel®
Drug: Zoledronic Acid — Phase I: First Cohort = 4 mg IV Over 15 min. every 4 Weeks; Next Cohort = Dose Expansion or Reduction Based on Dose Limiting Toxicity (DLT) in Initial Cohort.
  Phase II: Recommended Phase II Dose (RP2D) as determined with Phase I.
  Other Names: Zoledronate; Zometa®

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of dasatinib and Zometa (zoledronic acid) that can be given in combination for the treatment of breast cancer that has spread to the bone. The safety and effectiveness of this combination will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Zoledronic acid is designed to strengthen the bone and prevent fractures or breaks in the bone. Dasatinib is designed to block (stop) cells responsible for the breakdown of bone.

Study Groups:

If you are found to be eligible to take part in this study, you will be enrolled in a group of at least 3 participants to begin receiving zoledronic acid and dasatinib. The dose of dasatinib you receive will depend on when you enrolled in this study. All participants will receive the same amount of zoledronic acid. The first group of participants will be treated with the lowest dose of dasatinib given in combination with zoledronic acid.

Once the highest tolerable dose level is found, up to 25 additional participants will be enrolled at that dose level. This is called the Phase II portion of the study.

Drug Administration:

You will receive zoledronic acid through a needle in your vein on Day 1 over 15 minutes. You will take dasatinib by mouth daily for 28 days. Dasatinib should be taken on an empty stomach or after a light meal. Every 28 days is called a study "cycle."

Study Visits for Participants in the Phase I Portion:

On Day 1 of Cycle 1, you will have the following tests and procedures performed.

* You will have a physical exam, including measurement of your vital signs.
* You will have a performance status evaluation.
* Blood (about 1-2 teaspoons) will be drawn for routine tests.
* You will have an ECG.

On Day 8 of Cycle 1, you will have the following tests and procedures performed.

* Blood (about 1-2 teaspoons) will be drawn for routine tests.
* You will have an ECG.

On Day 15 of Cycle 1, you will have the following tests and procedures performed.

* You will have a physical exam.
* You will have a performance status evaluation.
* Blood (about 1-2 teaspoons) will be drawn for routine tests.
* You will have an ECG.

On Day 21 of Cycle 1, you will have the following tests and procedures performed.

* Your vital signs will be measured.
* Blood (about 1-2 teaspoons) will be drawn for routine tests.
* You will have an ECG.

On Day 1 of Cycle 2, you will have an ECG.

On Day 1 of all other cycles, you will have the following tests and procedures performed.

* You will have a physical exam.
* You will have a performance status evaluation.
* Blood (about 1-2 teaspoons) will be drawn for routine tests.
* You will have MRIs, CT scans, and/or x-rays to check the status of the disease.

On Days 1 and 28 of Cycle 1 and then every 3rd month, urine will be collected over 24 hours to check for markers of bone loss.

After Cycles 3, 6, 9 and so on, you will have CT scans, MRIs, and/or x-rays to check the status of the disease

At all study visits, you will be asked about any drugs you may be taking and any side effects you may be experiencing.

Study Visits for Participants in the Phase II Portion:

On Day 1 of all cycles, you will have the following tests and procedures performed.

* You will have a physical exam, including measurement of your vital signs.
* You will have a performance status evaluation.
* Blood (about 1-2 teaspoons) will be drawn for routine tests.

On Days 1 and 28 of Cycle 1 and then every 3rd month, urine will be collected to check for markers of bone loss.

After Cycles 2, 4, 6 and so on, you will have CT scans, MRIs, and/or x-rays to check the status of the disease.

At all study visits, you will be asked about any drugs you may be taking and any side effects you may be experiencing.

Length of Study:

You may remain on study for as long as you are benefitting. You will be taken off study if the disease gets worse or you experience intolerable side effects.

End-of-Study Visit:

Once you go off-study, you will have an end-of-study visit.

* Your vital signs will be measured.
* Blood (about 1-2 teaspoons) and urine will be collected for routine tests.
* You will have MRIs, CT scans, and/or x-rays to check the status of the disease.

This is an investigational study. Zoledronic acid is FDA approved and commercially available for the treatment of breast cancer. Dasatinib is not FDA approved or commercially available for the treatment of breast cancer. It has been authorized for use in research only. Up to 28 patients will take part in this multicenter study. Up to 12 will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a pathologically confirmed diagnosis of invasive carcinoma of the breast.
2. Patients must carry a diagnosis of metastatic breast cancer with predominant bone involvement. For the purposes of this study, predominant bone involvement will be defined as radiographically detected bone metastasis in the presence or absence of other sites of metastatic breast cancer (i.e. visceral involvement). If visceral involvement is present, patients must be asymptomatic and have no tumors in visceral organs that measure >3cm in size.
3. Patients must agree to serial urine collections for measurement of Ntx.
4. Age >/= 18 years.
5. Patients must be able to swallow oral medications. Dasatinib must be taken whole and cannot be crushed.
6. Patients must have evaluable disease using WHO Criteria for Assessment of Disease Response in Bone or MDACC Modified Response Criteria for Assessment of Disease Response in Bone.
7. Patients must not have had >1 chemotherapy regimens for metastatic disease. Patients with metastasis diagnosed </= 6 months after completion of adjuvant chemotherapy are considered to have had chemotherapy for metastatic breast cancer.
8. Patients with ER positive disease must have had disease progression on at least one prior hormonal therapy for metastatic disease. Patients must also have developed disease progression on their most recent hormonal therapy regimen and be agreeable to continue this regimen in combination with protocol therapy. For the purposes of this study disease progression while receiving hormonal therapy will be defined as: Radiographic evidence of progressive disease according to RECIST criteria, Progression of disease by physical exam in patients with skin involvement. Continued in # 9
9. Continuation from # 8: 25% increase in tumor marker as measured on two evaluations no less than 72 hours apart.
10. Patients must have and ECOG performance status of </= 2.
11. Patients must not require concurrent radiation or chemotherapy while receiving protocol therapy.
12. Patients must not have an active infection requiring the use of intravenous antibiotics. The use of oral antibiotics as prophylaxis is allowed.
13. Patients must have a baseline ECG with QTc within the normal range within 28 days prior to registration.
14. Patients must be informed of the investigational nature of the study and must sign and give written informed consent.
15. Patients may have received previous radiation but must have completed radiation at least 2 weeks (8 weeks for radiation to the brain) prior to registration. Patients with irradiated tumor as the only site of evaluable disease will not be eligible for protocol therapy unless there is documented disease progression within the previously radiated site.
16. Patients must have recovered to grade </= 1 from all acute toxicity of previous radiation or hormonal therapy.
17. Adequate hematologic and hepatic function: Granulocyte count >/= 1,500/mcL, Platelet count >/= 100,000/mcL, Bilirubin </= 1.5 x ULN, AST and/or ALT </= 2 x ULN, Alkaline phosphatase (liver component, if fractionated) </= 2 x ULN, Serum Na, K+, Mg2+, Phosphate and Ca2+>/= Lower Limit of Normal (LLN) [subjects with low electrolyte levels must be repleted to normal for protocol entry]
18. Patients must not receive any concurrent bisphosphonate therapy other than that prescribed by the study.
19. Sexually active patients with reproductive potential must agree to use an effective method of birth control during the course of the study and for no less than 4 weeks after discontinuing study drug. Contraceptives must be used in a manner such that risk of failure is minimized. Oral contraceptives should be avoided in women with estrogen or progesterone receptor positive breast cancer.
20. Prior to study enrollment, women of childbearing potential (WOCBP) must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy. In addition, men enrolled on this study should understand the risks to any sexual partner of childbearing potential and should practice an effective method of birth control.
21. All WOCBP MUST have a negative serum or urine pregnancy test within 72 hours prior to the start of study drug administration. If the pregnancy test is positive, the patient must not receive investigational product and must not be enrolled in the study.
22. Patients with disease progression while receiving previous therapy in combination with bisphosphonates (including zoledronic acid) will be considered eligible for protocol participation.

Exclusion Criteria:

1. Any malignancy (other than breast cancer) that required radiotherapy or systemic treatment within the past 5 years.
2. Concurrent medical condition which may increase the risk of toxicity, including: Pleural or pericardial effusion of any grade, clinically-significant coagulation or platelet function disorder (e.g. known von Willebrand's disease)
3. Cardiac Symptoms, including the following: Uncontrolled angina, congestive heart failure or MI within (6 months), diagnosed congenital long QT syndrome, any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes), prolonged QTc interval on pre-entry electrocardiogram (> normal range), subjects with hypokalemia or hypomagnesemia if it cannot be corrected
4. History of significant bleeding disorder unrelated to cancer, including: diagnosed congenital bleeding disorders (e.g., von Willebrand's disease), diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies), ongoing or recent (</= 3 months) significant gastrointestinal bleeding
5. Concomitant Medications, consider the following prohibitions (Drugs must be discontinued for 7 days prior to starting protocol therapy):
6. Women and men of child bearing potential: who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 4 weeks after cessation of study drug, or women of childbearing potential (CBP) who have a positive pregnancy test at baseline, or women who are pregnant or breastfeeding
7. Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious) illness
8. Untreated or uncontrolled brain metastasis
9. Patient inability to take or absorb oral medications
10. Current active dental problems including: ongoing infection of the teeth or jawbone (maxilla or mandibula); current exposed bone in the mouth; and current or prior diagnosis of osteonecrosis of the jaw
11. Recent (within 8 weeks) or planned dental or jaw surgery (e.g., extraction, implants)
12. Diagnosis of metabolic bone disease other than osteoporosis (e.g., Paget's disease of bone)
13. Known hypersensitivity to zoledronic acid or aspirin
14. Corrected serum calcium < 8.0 mg/dL (2.0 mmol/L) or >/= 12.0 mg/dL (3.0 mmol/L) at Visit 1. The formula to be used is: Corrected serum calcium (mg/dL) = Patient's serum calcium (mg/dL) + [0.8 x Midrange Albumin (g/dL) - Patient's Albumin (g/dL)]. 4.0g/dL to be used for the Midrange Albumin
15. Serum creatinine greater than or equal to 1.5 times the institutional upper limits of normal or a creatinine clearance of <40 ml/min when calculated by the Cockcroft and Gault formula (see protocol text for formula)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-11-01 (Actual); Primary Completion 2020-11-17 (Actual); Study Completion 2020-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacy Moulder, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - University of Chicago, Chicago, Illinois
  - Duke University, Durham, North Carolina
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled and treated on protocol at the three recruiting sites (MD Anderson Cancer, University of Chicago and Duke Cancer Institute).
Pre-assignment Details: 31 participants enrolled, 25 started treatment and 6 did not receive treatment.
Groups:
- Phase I Dasatinib (70 mg): Dasatinib 70 mg twice daily. Zoledronic acid was administered using standard dosing as a 15-minute intravenous infusion on day 1 of a 28-day cycle. Dasatinib was taken orally daily on days 1-28 of the cycle. Dasatinib was given continuously unless patients developed toxicities requiring dose adjustment or treatment interruption.
- Phase 1 Dasatinib (100 mg): Dasatinib (100 mg) daily. Zoledronic acid was administered using standard dosing as a 15-minute intravenous infusion on day 1 of a 28-day cycle. Dasatinib was taken orally daily on days 1-28 of the cycle. Dasatinib was given continuously unless patients developed toxicities requiring dose adjustment or treatment interruption.
- Phase II Drug Administration: Dasatinib 100 mg daily in combination with zoledronic acid 4 mg IV on day 1 of a 28-day cycle.
Period: Overall Study
Arm/Group | Phase I Dasatinib (70 mg) | Phase 1 Dasatinib (100 mg) | Phase II Drug Administration
Started | 1 | 6 | 18
Completed | 0 | 0 | 0
Not Completed | 1 | 6 | 18

BASELINE CHARACTERISTICS:
Population: Participants baseline characteristics are summarized due to the PI, Stacy Moulder, and those affiliated with the protocol is no longer at the institution. Baseline Data are combined based on the published article. We have attempted to the best of our ability to locate the Baseline Data per intervention for each phase but we were unsuccessful.
Groups:
- Phase I/Phase II: PhI/PhII- Dasatinib 70 mg twice daily/ dasatinib 100 mg daily in combination with zoledronic acid 4 mg IV on day 1 of a 28-day cycle.
Arm/Group | Phase I/Phase II
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 45 [36 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 25
Hormone Receptor [Count of Participants; unit: Participants]
  Positive | 21
  Negative | 4
Initial sites of metastases [Count of Participants; unit: Participants]
  Bone only | 17
  Lung | 5
  Lymph nodes | 4
  Liver | 1
Prior endocrine therapy for metastatic disease [Count of Participants; unit: Participants]
  0 | 7
  1 | 15
  >=2 | 3
Prior chemotherapy for metastatic disease [Count of Participants; unit: Participants]
  0 | 23
  1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response in Bone From Time of Initiation of Therapy to > 6 Months
Description: Objective response rate is defined as the clinical benefit rate (complete and partial response) + stable disease > 6 months in bone.
Time Frame: 6 months
Population: ITT, intent-to-treat analysis of all patients combined. The PI, Stacy Moulder, and those affiliated with the protocol is no longer at the institution. The objective response in bone from time to initiation of therapy to >6 months analysis are combined based on the published article. We have attempted to the best of our ability to locate the data for each phase but we were unsuccessful.
Measure: Count of Participants; unit: Participants
Groups:
- Phase I/Phase II: PhI/PhII-Open Label dasatinib 100 mg daily in combination with zoledronic acid 4 mg IV on day 1 of a 28-day cycle
Arm/Group | Phase I/Phase II
Number analyzed (Participants) | 25
Participants
  Central Review | 8
  Site Review | 7

2. Primary Outcome: Phase I - Maximum Tolerated Dose (MTD) and Recommended Phase II Dose (RP2D) for Dasatinib in Combination With Zoledronic Acid
Description: To determine the maximum tolerated dose (MTD) and recommended phase II dose (RP2D) for dasatinib in combination with zoledronic acid.
Time Frame: day 1 (+/- 48 hours) prior to therapy during cycle 2 and all subsequent cycles
Measure: Number; unit: mg
Groups:
- Phase I: Dasatinib 70 mg twice daily. Zoledronic acid was administered using standard dosing as a 15-minute intravenous infusion on day 1 of a 28-day cycle. Dasatinib was taken orally daily on days 1-28 of the cycle. Dasatinib was given continuously unless patients developed toxicities requiring dose adjustment or treatment interruption.
Arm/Group | Phase I
Number analyzed (Participants) | 7
mg
  Dasatinib | 100
  zoledronic acid | 4

ADVERSE EVENTS:
Time Frame: on day 1 (±48 hours) prior to therapy during subsequent cycles, up to 6 months
Description: The PI, Stacy Moulder, and those affiliated with the protocol is no longer at the institution. The adverse events are combined based on the published article. We have attempted to the best of our ability to locate the AEs for each phase but we were unsuccessful.
Arm/Group | Phase I/Phase II
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 9/25
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I/Phase II (N=25)
Anemia (Blood and lymphatic system disorders) | 3
Fatigue (General disorders) | 9
Rash (Skin and subcutaneous tissue disorders) | 9
Nausea (Gastrointestinal disorders) | 6
Pain (General disorders) | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Respiratory (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Vasomotor symptoms (Respiratory, thoracic and mediastinal disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 4
Diarrhea (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Xerostomia (General disorders) | 2
Vomiting (Gastrointestinal disorders) | 3
Infections (non-neutropenic) (Infections and infestations) | 3
Edema (Skin and subcutaneous tissue disorders) | 2
Paresthesia (Nervous system disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-03-28): https://cdn.clinicaltrials.gov/large-docs/18/NCT00566618/Prot_SAP_000.pdf